CLINICAL TRIAL: NCT03519763
Title: Endometrial and Isthmic Microbiota During IVF Stimulation in Patients Affected With Isthmocele and Intrauterine Mucus Secretion After C-section.
Brief Title: Intrauterine Microbiota During IVF in Patients Affected With Isthmocele.
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Prof Dr. Human Fatemi, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 1707-ABU-065-HF
Record Dates: First submitted 2018-04-25; First posted 2018-05-09 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Diseases
MeSH Terms: conditions — Uterine Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples for Endometrial fluid (EF) and isthmocele fluid (IF) will be collected the day of the oocyte pick up after IVF stimulation for freeze-all oocytes or embryos.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Fifteen patients without isthmocele
  Interventions: Diagnostic Test: ultrasound
- Study subgroup1: 15 patients with 1 previous C-Section
- Study subgroup2: 15 patients with 2 or more previous C-Section.
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — All the patients will have a transvaginal ultrasound evaluation during the first visit to the clinic to evaluate the presence or not of isthmocele.
  Other Names: transvaginal scan, ultrasound
  Groups: Control group; Study subgroup2

SUMMARY:
To evaluate the endometrial and isthmic microbiota in patients with isthmocele after C-Section, and if this microbiota is similar or not with better reproductive outcomes.

DETAILED DESCRIPTION:
A total of 45 subjects undergoing in vitro fertilization treatment. Fifteen patients without isthmocele will be included in the control group and 30 patients affected with isthmocele in the other group, divided in 2 subgroups: 15 with 1 previous C-Section, and 15 with 2 or more previous C-Section. Paired samples of endometrial fluid (EF) and isthmic fluid (IF) will be obtained simultaneously the day of egg retrieval. Patients will follow a protocol for all-freezing embryos or oocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with isthmocele:

   * Patients performing IVF treatment with a planned cycle segmentation and consecutive frozen embryo transfer on a hormone replacement therapy (HRT) cycle or natural cycle.
   * Age between 18 - 45 years all (both inclusive).
   * One or multiple C-sections.
   * Isthmocele present during TV scan.
   * BMI: 18,5 - 35 kg / m2 (both inclusive).
2. Patients without isthmocele:

   * Patients performing IVF treatment with planned cycle segmentation and who would have embryo transfer with frozen embryos under hormone replacement therapy.
   * NO Isthmocele present during transvaginal ultrasound.
   * BMI: 18,5 - 30 kg / m2 (both inclusive).

Exclusion Criteria:

* Age < 18 and > 45 years old.
* Previous or active endometritis.
* Patients who are IUD carriers for the last 3 months.
* Patients who have taken prescribed antibiotics in the last 3 months previous to sample collection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Female patients undergoing IVF treatment.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
If the intrauterine microbiota profile in patients affected with isthmocele differs from the one found in patients without isthmocele. | 1year
  patients undergoing in vitro fertilization treatment

CONTACTS AND LOCATIONS:
Overall Officials: Human Fatemi, MD, Principal Investigator — Medical Director
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sirota I, Zarek SM, Segars JH. Potential influence of the microbiome on infertility and assisted reproductive technology. Semin Reprod Med. 2014 Jan;32(1):35-42. doi: 10.1055/s-0033-1361821. Epub 2014 Jan 3. PMID 24390919
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Background] Romero R, Hassan SS, Gajer P, Tarca AL, Fadrosh DW, Bieda J, Chaemsaithong P, Miranda J, Chaiworapongsa T, Ravel J. The vaginal microbiota of pregnant women who subsequently have spontaneous preterm labor and delivery and those with a normal delivery at term. Microbiome. 2014 May 27;2:18. doi: 10.1186/2049-2618-2-18. eCollection 2014. PMID 24987521
- [Background] Moreno I, Codoner FM, Vilella F, Valbuena D, Martinez-Blanch JF, Jimenez-Almazan J, Alonso R, Alama P, Remohi J, Pellicer A, Ramon D, Simon C. Evidence that the endometrial microbiota has an effect on implantation success or failure. Am J Obstet Gynecol. 2016 Dec;215(6):684-703. doi: 10.1016/j.ajog.2016.09.075. Epub 2016 Oct 4. PMID 27717732
- [Background] Tower AM, Frishman GN. Cesarean scar defects: an underrecognized cause of abnormal uterine bleeding and other gynecologic complications. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):562-72. doi: 10.1016/j.jmig.2013.03.008. Epub 2013 May 14. PMID 23680518
- [Background] Vikhareva Osser O, Valentin L. Risk factors for incomplete healing of the uterine incision after caesarean section. BJOG. 2010 Aug;117(9):1119-26. doi: 10.1111/j.1471-0528.2010.02631.x. PMID 20604776
- [Background] Sim K, Cox MJ, Wopereis H, Martin R, Knol J, Li MS, Cookson WO, Moffatt MF, Kroll JS. Improved detection of bifidobacteria with optimised 16S rRNA-gene based pyrosequencing. PLoS One. 2012;7(3):e32543. doi: 10.1371/journal.pone.0032543. Epub 2012 Mar 28. PMID 22470420
- [Background] Caporaso JG, Kuczynski J, Stombaugh J, Bittinger K, Bushman FD, Costello EK, Fierer N, Pena AG, Goodrich JK, Gordon JI, Huttley GA, Kelley ST, Knights D, Koenig JE, Ley RE, Lozupone CA, McDonald D, Muegge BD, Pirrung M, Reeder J, Sevinsky JR, Turnbaugh PJ, Walters WA, Widmann J, Yatsunenko T, Zaneveld J, Knight R. QIIME allows analysis of high-throughput community sequencing data. Nat Methods. 2010 May;7(5):335-6. doi: 10.1038/nmeth.f.303. Epub 2010 Apr 11. No abstract available. PMID 20383131